CLINICAL TRIAL: NCT00616421
Title: A Phase 3, Randomized, Observer-blind, Multi-Center Study to Compare the Safety and Immunogenicity of One Dose of Novartis Meningococcal ACWY Conjugate Vaccine With One Dose of Licensed Meningococcal ACWY Conjugate Vaccine Administered to Healthy Children 2-10 Years of Age
Brief Title: Safety and Immune Response of Novartis of MenACWY Conjugate Vaccine When Given to Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V59P20; 11278
Record Dates: First submitted 2008-01-31; First posted 2008-02-15 (Estimated); Results first posted 2011-06-09 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Meningococcal Infections
Keywords: vaccine; children; healthy; meningitis; meningococcal; prevention of meningococcal disease serogroups ACWY; Menveo
MeSH Terms: conditions — Meningococcal Infections; Meningitis | interventions — MenACWY-CRM vaccine; Meningococcal Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MenACWY-CRM (1 dose) (Experimental): 1 injection of the Novartis MenACWY-CRM (a nontoxic mutant of diptheria toxin) conjugate vaccine administered by intramuscular (IM) injection on study day 1.
  Interventions: Biological: MenACWY-CRM
- Licensed polysaccharide vaccine (Active Comparator): 1 injection of a licensed meningococcal MenACWY polysaccharide-protein conjugate vaccine administered by intramuscular (IM) injection on study day 1
  Interventions: Biological: Licensed meningococcal ACWY vaccine
- MenACWY-CRM (2 doses) (Experimental): 2 injections of the Novartis MenACWY-CRM (a nontoxic mutant of diptheria toxin) conjugate vaccine administered by intramuscular (IM) injection on study days 1 and 61.
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM — 1 injection of the Novartis MenACWY-CRM conjugate vaccine administered intramuscularly
  Other Names: Menveo
  Arms: MenACWY-CRM (1 dose)
Biological: MenACWY-CRM — 2 injections of the Novartis MenACWY-CRM conjugate vaccine administered intramuscularly to children 2 to 5 years of age
  Other Names: Menveo
  Arms: MenACWY-CRM (2 doses)
Biological: Licensed meningococcal ACWY vaccine — 1 injection of the licensed meningococcal ACWY was administered intramuscularly
  Other Names: Menactra
  Arms: Licensed polysaccharide vaccine

SUMMARY:
To evaluate the safety and immune response of Novartis MenACWY conjugate vaccine when given to healthy children compared to a licensed Meningococcal ACWY polysaccharide-protein conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

* healthy 2-10 years of age children, inclusive and for whom, after the nature of the study has been explained, the parent or legal guardian has provided written informed consent
* who are available for all visits and telephone calls scheduled for the study
* who are up-to-date with age-appropriate routine childhood vaccinations

Exclusion Criteria:

* whose parent or legal guardian is unwilling or unable to give written informed consent
* who had a previous or suspected disease caused by N. meningitidis;
* who have previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s)
* who have received any investigational agents or vaccines within 90 days prior to enrollment
* who have any serious acute, chronic or progressive disease
* who have epilepsy or any progressive neurological disease or history of Guillain Barré Syndrome
* who have a history of anaphylaxis, serious vaccine reactions
* who have a known or suspected impairment/alteration of immune function, either congenital or acquired or resulting from
* who are known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time
* who have Down's syndrome or other known cytogenic disorders

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2907 (Actual)
Dates: Start 2008-03; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (63):
- United States (48):
  - Children's Investigational Reserach Program, Bentonville, Arkansas
  - Arkansas Pediatric Research Group, Little Rock, Arkansas
  - Premier Health Research Center, Downey, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente - Fresno, Fresno, California
  - Kaiser Permanente - Hayward, Hayward, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Kaiser Permanente - Pleasanton, Pleasanton, California
  - Kaiser Permanente - San Francisco, San Francisco, California
  - Kaiser Permanente - San Jose, San Jose, California
  - Kaiser Permanente - Aurora, Aurora, Colorado
  - 1st Allergy & Clinical Research, Centennial, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - 1st Allergy & Clinical Research, Thornton, Colorado
  - Kaiser Permanente - Westminister, Westminister, Colorado
  - Kentucky Pediatric Research Center, Bardstown, Kentucky
  - Physicians to Children & Adolescents, Springfield, Kentucky
  - Benchmark Research, Metairie, Louisiana
  - St. Louis University School of Medicine, St Louis, Missouri
  - Meridian Clinical Research LLC, Omaha, Nebraska
  - Legacy Pediatrics, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Durham Pediatrics, Durham, North Carolina
  - Regional Pediatric Associates PA, Durham, North Carolina
  - Odyssey Research, Fargo, North Dakota
  - Dr. Senders and Associates, Cleveland, Ohio
  - Calcagno Research & Development, Gresham, Oregon
  - Children's Health Care - West, Erie, Pennsylvania
  - University Of Pittsburgh Medical Center, Greenville, Pennsylvania
  - Family Healthcare Partners, Grove City, Pennsylvania
  - Pediatric Associates of Latrobe, Latrobe, Pennsylvania
  - Pediatric Alliance PC, Pittsburgh, Pennsylvania
  - South Hills Pediatrics, Pittsburgh, Pennsylvania
  - Primary Physicians Research Inc., Pittsburgh, Pennsylvania
  - Laurel Pediatrics, Uniontown, Pennsylvania
  - Family Practice Medical Associates South, Upper Saint Clair, Pennsylvania
  - Children's Community Pediatrics, Wexford, Pennsylvania
  - Jackson Clinic Professional Association, Jackson, Tennessee
  - Benchmark Research Ft. Worth, Fort Worth, Texas
  - Benchmark Research San Angelo, San Angelo, Texas
  - Jean Brown Research, Clinton, Utah
  - Wee Care Pediatrics, Layton, Utah
  - Cottonwood Pediatrics, Murray, Utah
  - J. Lewis Research Inc., Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Copperview Medical Center, South Jordan, Utah
  - Rockwood Clinic, Spokane, Washington
  - Rockwood Clinic North, Spokane, Washington
- Canada (15):
  - TASC Research Services Inc., Surrey, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Clinical Trials Research Center, Halifax, Nova Scotia
  - Colchester Regional Hospital, Truro, Nova Scotia
  - Albion Finch Medical Centre, Etobicoke, Ontario
  - Medicor Research Inc., Greater Sudbury, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - SKDS Research In., Newmarket, Ontario
  - Herridge Community Health Clinic, Ottawa, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Resolve Research Solutions, Toronto, Ontario
  - Queen Elizabeth Hospital, Charlottetown, Prince Edward Island
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Commonwealth Medical Clinic, Mount Pearl
  - White Hills Medical Clinic, St. John's

REFERENCES:
- [Result] Halperin SA, Gupta A, Jeanfreau R, Klein NP, Reisinger K, Walter E, Bedell L, Gill C, Dull PM. Comparison of the safety and immunogenicity of an investigational and a licensed quadrivalent meningococcal conjugate vaccine in children 2-10 years of age. Vaccine. 2010 Nov 23;28(50):7865-72. doi: 10.1016/j.vaccine.2010.09.092. Epub 2010 Oct 29. PMID 20943209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 67 centers in the USA and Canada.
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- MenACWY-CRM (2 Doses): 2 injections of the Novartis MenACWY-CRM (a nontoxic mutant of diptheria toxin) vaccine administered by intramuscular (IM) injection on study days 1 and 61 in children 2 to 5 years of age
- MenACWY-CRM (1 Dose): 1 injection of the Novartis MenACWY-CRM (a nontoxic mutant of diptheria toxin) vaccine administered by intramuscular (IM) injection on study day 1
- Licensed Polysaccharide Vaccine: 1 injection of the licensed meningococcal MenACWY polysaccharide vaccine administered on study day 1
Period: Overall Study
Arm/Group | MenACWY-CRM (2 Doses) | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine
Started | 359 | 1278 | 1270
Completed | 333 | 1240 | 1229
Not Completed | 26 | 38 | 41
Not completed — Withdrawal by Subject | 9 | 11 | 8
Not completed — Lost to Follow-up | 12 | 26 | 30
Not completed — Inappropriate enrollment | 3 | 0 | 1
Not completed — Administrative reason | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 2
Not completed — Unable to classify | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MenACWY-CRM (2 Doses): 2 injections of the Novartis MenACWY-CRM vaccine administered on study days 1 and 61 in children 2 to 5 years of age.
- MenACWY-CRM (1 Dose): 1 injection of the Novartis MenACWY-CRM (a nontoxic mutant of diptheria toxin) vaccine administered by intramuscular (IM) injection on study day1.
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM (2 Doses) | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine | Total
Number analyzed (Participants) | 359 | 1278 | 1270 | 2907
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.5 (1.1) | 5.5 (2.5) | 5.6 (2.6) | 5.3 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 622 | 580 | 1373
  Male | 188 | 656 | 690 | 1534

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With hSBA Seroresponse, in Healthy Children 2 to 5 Years of Age
Description: The immunogenicity of a single dose of MenACWY-CRM is compared with the immunogenicity of a single dose of the licensed ACWY polysaccharide vaccine, in terms of the percentages of subjects with seroresponse directed against N. meningitidis serogroups A, C, W-135, and Y.
  Seroresponse: For a subject with hSBA <1:4 at baseline, seroresponse is defined as a postvaccination hSBA ≥ 1:8; for a subject with hSBA ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM (1 Dose): 1 injection of the Novartis MenACWY-CRM (a nontoxic diptheria toxin) vaccine administered on study day 1
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 607 | 615
Percentages of subjects
  Serogroup A (N=606, 611) | 72 [68 to 75] | 77 [73 to 80]
  Serogroup C (N=607, 615) | 60 [56 to 64] | 56 [52 to 60]
  Serogroup W (N=594, 605) | 72 [68 to 75] | 58 [54 to 62]
  Serogroup Y (N=593, 600) | 66 [62 to 70] | 45 [41 to 49]

2. Secondary Outcome: Percentages of Subjects With hSBA Seroresponse, in Healthy Children 2 to 10 Years of Age.
Description: as for outcome 1
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percenatage of subjects
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 1161 | 1154
Percenatage of subjects
  Serogroup A (N=1157, 1152) | 74 [71 to 76] | 80 [77 to 82]
  Serogroup C (N=1161, 1154) | 61 [58 to 64] | 57 [54 to 60]
  Serogroup W (N=1136, 1138) | 65 [62 to 67] | 51 [48 to 54]
  Serogroup Y (N=1138, 1139) | 62 [60 to 65] | 42 [40 to 45]

3. Primary Outcome: Percentages of Subjects With hSBA Seroresponse, in Healthy Children 6 to 10 Years of Age.
Description: The immunogenicity of a single dose of MenACWY-CRM is compared with the immunogenicity of a single dose of the licensed ACWY polysaccharide vaccine, in terms of the percenatages of subjects with seroresponse directed against N. meningitidis serogroups A, C, W-135, and Y.
  Seroresponse: For a subject with hSBA <1:4 at baseline, seroresponse is defined as a postvaccination hSBA ≥ 1:8; for a subject with hSBA ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 554 | 541
Percentages of subjects
  Serogroup A (N=551, 541) | 77 [73 to 80] | 83 [79 to 86]
  Serogroup C (N=554, 539) | 63 [59 to 67] | 57 [53 to 62]
  Serogroup W (N=542, 533) | 57 [53 to 61] | 44 [40 to 49]
  Serogroup Y (N=545, 539) | 58 [54 to 62] | 39 [35 to 44]

4. Secondary Outcome: Percentages of Subjects With hSBA ≥ 1:8, in Healthy Children 2 to 10 Years of Age
Description: as for outcome 1
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 1161 | 1154
Percentage of subjects
  Serogroup A (N=1157, 1152) | 75 [72 to 77] | 80 [78 to 83]
  Serogroup C (N=1161, 1154) | 72 [70 to 75] | 68 [66 to 71]
  Serogroup W (N=1136, 1138) | 90 [88 to 92] | 60 [57 to 63]
  Serogroup Y (N=1138, 1139) | 77 [75 to 80] | 79 [77 to 81]

5. Secondary Outcome: Geometric Mean Titers (hSBA), in Healthy Children 2 to 10 Years of Age.
Description: The immunogenicity of a single dose of MenACWY-CRM is compared with the immunogenicity of a single dose of the licensed ACWY polysaccharide vaccine, in terms of the number of subjects with hSBA (human Serum Bactericidal Activity) Geometric Mean Titers (GMTs) response against N. meningitidis serogroups A, C, W-135, and Y.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 1161 | 1154
Titers
  Serogroup A (N=1157, 1152) | 30 [27 to 31] | 29 [26 to 33]
  Serogroup C (N=1161, 1154) | 23 [21 to 27] | 17 [15 to 20]
  Serogroup W (N=1136, 1138) | 49 [44 to 54] | 26 [23 to 29]
  Serogroup Y (N=1138, 1139) | 29 [25 to 32] | 12 [11 to 14]

6. Secondary Outcome: Percentages of Subjects With hSBA ≥ 1:8, in Healthy Children 2 to 5 and 6 to 10 Years of Age.
Description: The immunogenicity of a single dose of MenACWY-CRM is compared with the immunogenicity of a single dose of the licensed ACWY polysaccharide vaccine, in terms of the percenategs of subjects with seroresponse directed against N. meningitidis serogroups A, C, W-135, and Y.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM (2 to 5 Yoa): 1 injection of the Novartis MenACWY-CRM vaccine administered by IM on study day 1 in children 2 to 5 years of age.
- Licensed Polysaccharide Vaccine (2 to 5 Yoa): 1 injection of the licensed meningococcal MenACWY polysaccharide vaccine administered by IM on study day 1 in children 2 to 5 years of age.
- MenACWY-CRM (6 to 10 Yoa): 1 injection of the Novartis MenACWY-CRM vaccine administered by IM on study day 1 in children 6 to 10 years of age.
- Licensed Polysaccharide Vaccine (6 to 10 Yoa): 1 injection of the licensed meningococcal ACWY polysaccharide-protein conjugate administered by IM on study day 1 in children 6 to 10 years of age.
Arm/Group | MenACWY-CRM (2 to 5 Yoa) | Licensed Polysaccharide Vaccine (2 to 5 Yoa) | MenACWY-CRM (6 to 10 Yoa) | Licensed Polysaccharide Vaccine (6 to 10 Yoa)
Number analyzed (Participants) | 607 | 554 | 615 | 541
Percentages of subjects
  Serogroup A (N=606, 611, 551, 541) | 72 [68 to 75] | 78 [74 to 81] | 77 [74 to 81] | 83 [80 to 86]
  Serogroup C (N=607, 615, 554, 539) | 68 [64 to 72] | 64 [60 to 68] | 77 [73 to 89] | 74 [70 to 77]
  Serogroup W (N=594, 605, 542, 533) | 90 [87 to 92] | 75 [71 to 78] | 91 [88 to 93] | 84 [81 to 87]
  Serogroup Y (N=593, 600, 545, 539) | 76 [72 to 79] | 57 [53 to 61] | 79 [76 to 83] | 63 [59 to 67]

7. Secondary Outcome: Geometric Mean Titers (hSBA), in Healthy Children 2 to 5 and 6 to 10 Years of Age.
Description: The immunogenicity of a single dose of the Novartis MenACWY-CRM is compared with the immunogenicity of a single dose of the licensed ACWY polysaccharide vaccine, in terms of the number of subjects with hSBA (human Serum Bacterial Activity) Geometric Mean Titers (GMTs) response against N. meningitidis serogroups A, C, W-135, and Y.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Licensed Polysaccharide Vaccine (6 to 10 Yoa): 1 injection of the licensed meningococcal MenACWY polysaccharide vaccine administered by IM on study day 1 in children 6 to 10 years of age
Arm/Group | MenACWY-CRM (2 to 5 Yoa) | Licensed Polysaccharide Vaccine (2 to 5 Yoa) | MenACWY-CRM (6 to 10 Yoa) | Licensed Polysaccharide Vaccine (6 to 10 Yoa)
Number analyzed (Participants) | 607 | 615 | 551 | 541
Titers
  Serogroup A (N=606, 611, 551, 541) | 26 [22 to 30] | 25 [21 to 29] | 35 [29 to 42] | 35 [29 to 41]
  Serogroup C (N=607, 615, 554, 539) | 18 [15 to 20] | 13 [11 to 15] | 36 [29 to 42] | 27 [21 to 33]
  Serogroup W (N=594, 605, 542, 533) | 43 [38 to 50] | 21 [19 to 25] | 61 [52 to 72] | 35 [30 to 42]
  Serogroup Y (N=593, 600, 545, 539) | 24 [20 to 28] | 10 [8.68 to 12] | 34 [28 to 41] | 14 [12 to 17]

8. Secondary Outcome: Percentages of Subjects With hSBA Seroresponse, in Healthy Children 2 to 5 Years of Age (2 Doses vs 1 Dose)
Description: The immunogenicity of two doses of the Novartis MenACWY-CRM, administered 2 months apart, is compared with the immunogenicity of a single dose of the Novartis MenACWY-CRM, directed against N. meningitidis serogroups A, C, W-135, and Y.
  Seroresponse: For a subject with hSBA <1:4 at baseline, seroresponse is defined as a postvaccination hSBA ≥ 1:8; for a subject with hSBA ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM (2 Doses): 2 injections of the Novartis MenACWY-CRM vaccine administered by IM on study days 1 and 61 in children 2 to 5 years of age
- MenACWY-CRM (1 Dose): 1 injection of the Novartis MenACWY-CRM vaccine administered by IM on study day 1 in children 2 to 5 years of age
Arm/Group | MenACWY-CRM (2 Doses) | MenACWY-CRM (1 Dose)
Number analyzed (Participants) | 293 | 607
Percentages of subjects
  Serogroup A (N=291, 606) | 91 [87 to 94] | 72 [68 to 75]
  Serogroup C (N=293, 607) | 98 [95 to 99] | 60 [56 to 64]
  Serogroup W (N=288, 594) | 89 [85 to 92] | 72 [68 to 75]
  Serogroup Y (N=286, 593) | 95 [91 to 97] | 66 [62 to 70]

9. Secondary Outcome: Percentages of Subjects With hSBA ≥ 1:8, in Healthy Children 2 to 5 Years of Age (2 Doses v/s 1 Dose)
Description: as for outcome 8
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM (2 Doses) | MenACWY-CRM (1 Dose)
Number analyzed (Participants) | 293 | 607
Percentages of subjects
  Serogroup A (N=291, 606) | 91 [88 to 94] | 72 [68 to 75]
  Serogroup C (N=293, 607) | 99 [97 to 100] | 68 [64 to 72]
  Serogroup W (N=288, 594) | 99 [98 to 100] | 90 [87 to 92]
  Serogroup Y (N=286, 593) | 98 [95 to 99] | 76 [72 to 79]

10. Secondary Outcome: GMTs (hSBA) in Healthy Children 2 to 5 Years of Age (2 Doses v/s 1 Dose)
Description: The immunogenicity of two doses of the Novartis MenACWY-CRM vaccine, administered 2 months apart, is compared with the immunogenicity of a single dose of the Novartis MenACWY-CRM vaccine, in terms of hSBA (human Serum Bactericidal Activity) GMTs (Geometric Mean Titers) against N. meningitidis serogroups A, C, W-135, and Y.
  ANOVA model used for the analysis of this outcome is different compare to ANOVA model used for the other outcome. The computed model components vary according to the variance observed due to the different datasets.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM (2 Doses) | MenACWY-CRM (1 Dose)
Number analyzed (Participants) | 293 | 607
Titers
  Serogroup A (N=291, 606) | 64 [51 to 81] | 27 [23 to 82]
  Serogroup C (N=293, 607) | 144 [118 to 177] | 18 [15 to 21]
  Serogroup W (N=288, 594) | 132 [111 to 157] | 41 [36 to 47]
  Serogroup Y (N=286, 593) | 102 [82 to 126] | 23 [20 to 27]

11. Secondary Outcome: Percentages of Subjects With at Least One Reactogenicity Sign After Vaccination in Children 2 to 5 Years of Age - 1 Dose Vaccine Treatment.
Description: Safety was assessed in terms of the percentages of subjects with reported local and systemic reactions up to 7 days after each vaccination per vaccination group, after 1 dose treatment.
Time Frame: Study days 1 to 7
Population: The analysis was performed on the safety population. Only groups receiving 1 dose vaccine are reported.
Measure: Number; unit: Percentages of subjects
Groups:
- MenACWY-CRM (1 Dose): The Novartis MenACWY-CRM vaccine was administered by IM in children 2 to 5 years of age.
- Licensed Polysaccharide Vaccine (1 Dose): The licensed meningococcal MenACWY polysaccharide vaccine was administered by IM in children 2 to 5 years of age.
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine (1 Dose)
Number analyzed (Participants) | 693 | 684
Percentages of subjects
  Injection site pain | 33 | 35
  Injection site erythema | 27 | 18
  Injection site induration | 18 | 18
  Change in Eating Habits (N=683, 671) | 9 | 10
  Sleepiness (N=692, 684) | 16 | 18
  Irritability (N=692, 684) | 21 | 22
  Vomiting (N=692, 684) | 3 | 3
  Diarrhea (N=692, 684) | 7 | 8
  Arthralgia | 3 | 4
  Headache | 5 | 6
  Rash | 4 | 5
  Fever ( ≥ 38C ; N=692, 684) | 2 | 2
  Fever ( ≥ 40.0C ) | 0 | 0
  Stayed home (N=682, 670) | 3 | 2
  Analgesic/Antipyretic medication used | 11 | 13

12. Secondary Outcome: Percentages of Subjects With at Least One Reactogenicity Sign After Vaccination in Children 6 to 10 Years of Age - 1 Dose Vaccine Treatment.
Description: Safety was assessed in terms of the percentages of subjects with reported local and systemic reactions up to 7 days after each vaccination per vaccination group after 1 dose treatment.
Time Frame: Study days 1 to 7
Population: The analysis was performed on the safety population. Only groups receiving 1 dose vaccine are reported.
Measure: Number; unit: Percenatage of subjects
Groups:
- MenACWY-CRM (1 Dose): The Novartis MenACWY-CRM vaccine was administered by IM in children 6 to 10 years of age.
- Licensed Polysaccharide Vaccine (1 Dose): The licensed meningococcal MenACWY polysaccharide vaccine was administered by IM in children 6 to 10 years of age.
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine (1 Dose)
Number analyzed (Participants) | 582 | 571
Percenatage of subjects
  Injection site pain | 39 | 45
  Injection site erythema | 28 | 22
  Injection site induration | 17 | 13
  Chills | 5 | 5
  Nausea | 8 | 6
  Malaise | 14 | 11
  Myalgia | 10 | 10
  Arthralgia | 6 | 4
  Headache | 18 | 13
  Rash | 5 | 3
  Fever ( ≥ 38C ; N=582, 570) | 2 | 2
  Fever ( ≥ 40.0C ; N=582, 570) | 0 | 1
  Stayed home (N=575, 566) | 3 | 2
  Analgesic/Antipyretic medication used | 9 | 10

13. Secondary Outcome: Percentages of Subjects With Unsolicited AEs Occurring Throughout the Study in Children Aged 2 to 10 Years - 1 Dose Vaccine Treatment.
Description: Safety was assessed in terms of the percentage of subjects with unsolicited AEs occurring throughout the entire study period, after 1 dose treatment.
Time Frame: day 1 to study termination (day 240)
Population: The analysis was performed on safety population. Only groups receiving 1 dose vaccine are reported.
Measure: Number; unit: Percentage of Subjects
Groups:
- Licensed Polysaccharide Vaccine (1 Dose): 1 injection of the licensed meningococcal MenACWY polysaccharide vaccine administered on study day 1
Arm/Group | MenACWY-CRM (1 Dose) | Licensed Polysaccharide Vaccine (1 Dose)
Number analyzed (Participants) | 1275 | 1255
Percentage of Subjects
  Any AEs | 26 | 24
  Possibly probably related AEs | 5 | 5
  SAEs | 1 | 1
  AEs leading to discontinuation | 0 | 0
  Possibly probably related SAEs | 0 | 0
  Death | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse events and serious adverse events were collectedfrom day 1 to study terminaton (day 240).
Description: If the adverse event was solicited then the event is listed as systematic assessment. However, if the adverse event was not solicited (i.e., unsolicited), then the event is listed under non-systematic method of collection. Subjects not vaccinated were excluded from the safety analysis.
Groups:
- MenACWY-CRM (1 Dose)_2 to 5 Years: 1 injection of the Novartis MenACWY-CRM vaccine administered on study day 1 in children 2 to 5 years of age.
- MenACWY-CRM (1 Dose)_6 to 10 Years: 1 injection of the Novartis MenACWY-CRM vaccine administered on study day 1 in children 6 to 10 years of age.
- Licensed Polysaccharide Vaccine_2 to 5 Years: 1 injection of the licensed meningococcal MenACWY polysaccharide vaccine administered on study day 1 in children 2 to 5 years of age.
- Licensed Polysaccharide Vaccine_6 to 10 Years: 1 injection of the licensed meningococcal MenACWY polysaccharide vaccine administered on study day 1 in children 6 to 10 years of age.
Arm/Group | MenACWY-CRM (2 Doses) | MenACWY-CRM (1 Dose)_2 to 5 Years | MenACWY-CRM (1 Dose)_6 to 10 Years | Licensed Polysaccharide Vaccine_2 to 5 Years | Licensed Polysaccharide Vaccine_6 to 10 Years
Serious Adverse Events (participants affected / at risk) | 2/351 | 5/693 | 3/582 | 5/684 | 2/571
Other Adverse Events (participants affected / at risk) | 253/351 | 424/693 | 340/582 | 419/684 | 342/571
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MenACWY-CRM (2 Doses) (N=351) | MenACWY-CRM (1 Dose)_2 to 5 Years (N=693) | MenACWY-CRM (1 Dose)_6 to 10 Years (N=582) | Licensed Polysaccharide Vaccine_2 to 5 Years (N=684) | Licensed Polysaccharide Vaccine_6 to 10 Years (N=571)
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth Cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Parvovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Peritonsillar Abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 1 | 0
Shigella infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis Staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Adrenal Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Pulmonary Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Loss of Consciousness (Nervous system disorders) | 0 (0) | 0 | 1 | 0 | 0
Psychiatric Symptom (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Bronchial Spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM (2 Doses) (N=351) | MenACWY-CRM (1 Dose)_2 to 5 Years (N=693) | MenACWY-CRM (1 Dose)_6 to 10 Years (N=582) | Licensed Polysaccharide Vaccine_2 to 5 Years (N=684) | Licensed Polysaccharide Vaccine_6 to 10 Years (N=571)
upper respiratory tract infection (Infections and infestations) | 20 | 13 | 4 | 9 | 1
injection site pain (General disorders) | 151 | 226 | 226 | 241 | 256
injection site erythema (General disorders) | 131 | 186 | 164 | 170 | 126
irritablility (General disorders) | 98 | 147 | 0 | 152 | 0
injection site induration (General disorders) | 82 | 126 | 97 | 126 | 73
somnolence (Nervous system disorders) | 81 | 109 | 0 | 126 | 0
headache (Nervous system disorders) | 27 | 37 | 105 | 39 | 79
mailaise (General disorders) | 0 | 0 | 82 | 0 | 62
eating disorder (Psychiatric disorders) | 56 | 64 | 0 | 69 | 0
diarrhoea (Gastrointestinal disorders) | 35 | 52 | 4 | 55 | 2
rash (General disorders) | 31 | 33 | 28 | 35 | 21
arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 25 | 38 | 24 | 25
pyrexia (General disorders) | 20 | 25 | 15 | 20 | 13
NAUSEA (Gastrointestinal disorders) | 3 | 2 | 50 | 0 | 37
VOMITING (Gastrointestinal disorders) | 19 | 25 | 2 | 22 | 5
CHILLS (General disorders) | 0 | 0 | 30 | 0 | 26
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 62 | 0 | 59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No